CLINICAL TRIAL: NCT00571792
Title: Evaluation of Airway Gene Expression in COPD and Controlled Populations
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: University of Nebraska (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0406-05-FB
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic testing involves identification of potential proteins and biomarkers produced from the DNA and RNA analysis. Included are MMP12 and MMP9, Nrf-2 gene, heme oxygenases, glutathione, sythesizing enzymes, thioredoxin reductase, NADPH dependent quinone reductase 1 as well as certain p450 members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- methodologies to identify characteristics of non-smokers with normal lung function: Imaging, genomic and proteomic methodologies to identify characteristics of individuals with normal lung function who do not smoke
- methodologies to identify characteristics of smokers but do not demonstrate symptoms of COPD: Imaging, genomic and proteomic methodologies to identify characteristics of individuals who smoke but who do not demonstrate symptoms of chronic obstructive pulmonary disease
- methodologies to identify characteristics of smokers that demonstrate symptoms of COPD: Imaging, genomic and proteomic methodologies to identify characteristics of individuals who smoke that demonstrate symptoms of COPD

SUMMARY:
To explore potential proteins that may be used to develop novel therapies for COPD. This will be accomplished by acquiring material from the lower respiratory tract via endobronchial brushings.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease(COPD) is currently the fourth leading cause of death in the United States. COPD is characterized by reduced airflow that is largely irreversible and progressive. Smoking is recognized as the most important cause of COPD contributing up to 80% of the cases. The disease does demonstrate a significant variability in airflow obstruction during the progression of the disease among those who are diagnosed and treated. This is probably due not only to the role of exposure of cigarette smoke and other noxious inhaled particles and gases but also to the individual's varied responses to those exposures.

COPD is characterized by an inflammatory response that does have a number of components that may be present in variable amounts. Recent data suggests that the cigarette exposure may cause several distinct pathophysiological processes that in turn may account for the variability demonstrated in altered lung structure that leads to functional impairment. Current therapies can help with alleviation of symptoms in individuals but not the unaltered course of loss in lung function that frequently leads to respiratory failure and death.

New strategies have been discussed as a means to new therapeutic approaches to altering the course of the disease. The use of genomic and proteomic methodologies offer promise to identify the pathways critical and relevant to the progression of COPD. To date approved medications target only the inflammatory response to the disease.

The study will explore metabolic pathways that could affect the remodeling process associated with the disease. Because of the heterogeneity of COPD, characteristics of the individual as well as between individuals must be identified in more detail. Mechanisms that enable this not only include physiological characterization by the current prescribed interventions but also imaging data which provides such ability to quantify airway wall thickness as well as via DNA that will be collected and save in order to gain a better understanding between the methodologies as they relate to the characterization of COPD. Currently, there may be a common understanding of how a particular drug affects a detailed molecular mechanism, however frequently it is not known why. The purpose of this study is to assist in discovery of the why.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-70 yrs of age, incl, women as described above as far as child-bearing potential and subjects who if they have coexisting disease, the disease is stable and does not place an untoward risk or result in compromise of data.
* Non smokers will be lifelong and have not worked in a chronic dusty environment.
* Smokers will require a minimum of 10 pkyr history and currently smoking at least a pack per day. The smokers without symptoms of COPD must demonstrate a pulmonary function with an FEV1 > 80%. The FEV1/FVC ratio may be less than .7 however they can not demonstrate symptoms of chronic bronchitis by medical history. Smokers with symptoms must demonstrate an FEV1 < 80% and FEV1/FVC <.7.

Exclusion Criteria:

* Any female subject who is pregnant or breast-feeding or a female subject who is of child-bearing potential who is unwilling to sue two acceptable methods of birth control.
* Any condition that would place the subject at risk for endobronchial brushings(such as bleeding diathesis) or subjects who are currently taking anticoagulants.
* Any subject who has had an exacerbation of COPD within the last six months of screening or who has been hospitalized for any reason within the last three months.
* Illicit substances indicated by positive urine drug screen.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males or non-pregnant, non-nursing females who are of non-childbearing potential between the ages of 45 and 70 years of age and who may be either life long non smokers, smokers who do not demonstrate symptoms of COPD and smokers who do demonstrate symptoms of COPD
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I Rennard, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States